CLINICAL TRIAL: NCT06886334
Title: Comparison of the Effects of Conventional Physical Therapy and Flexion-Distraction Technique on Pain, Functional Capacity, Activities of Daily Living, and Range of Motion in Patients with Lumbar Disc Herniation: a Randomized Controlled Trial
Brief Title: Flexion-Distraction Technique
Acronym: FDT
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gulay karacaoglu, Assistant Professor, Head of Physiotherapy and Rehabilitation Department, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-7694
Record Dates: First submitted 2025-03-07; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Lumbar Disc Herniation
Keywords: Pain; Range of Motion; Flexion-Distraction Technique; Conventional Physical Therapy
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 1. Conventional Physical Therapy Group (CTG): Ultrasound (4 minutes), TENS (100 Hz, 20 minutes), heat application (15 minutes), and home exercises will be applied. Treatment will be conducted three times a week for four weeks.
  2. Flexion-Distraction Group (Cox Technique) (CTG): In addition to heat application (15 minutes) and home exercises, the Cox technique will be used. The patient will be placed face down on a specialized table, and traction will be applied to the lumbar spine for 10 minutes.
Who Masked: Participant
Masking Description: Participants will be assigned in a blinded manner based on their preferred treatment center. Each center will administer a specific treatment protocol: one center will apply the flexion-distraction technique (Cox technique), while the other will provide conventional physical therapy. Participants will receive the treatment corresponding to the center they choose, ensuring that the allocation is based on their preference while maintaining the integrity of the study design. This approach allows for a natural randomization process while minimizing bias, as participants are unaware of the differences in treatment protocols between the centers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Physical Therapy Group (CPTG) (Active Comparator): A treatment protocol of ultrasound, TENS, hot pack, and exercises will be applied 3 times weekly for 4 weeks. Ultrasound (4 minutes per side) uses high-frequency waves for deep tissue healing. TENS (100 Hz, 20 minutes) delivers electrical currents to block pain signals. Hot packs (15 minutes) increase circulation and relax muscles. Exercises include Pelvic Tilt, Hip Flexor Stretch, Hamstring Stretch, Cat-Camel, Bridge, and Straight Leg Raise, aimed at improving flexibility, strength, and pain relief.
  Interventions: Other: exercise
- Flexion-Distraction Group (Cox Technique) (CTG): (Experimental): n addition to hot packs (15 minutes) and exercises, the flexion-distraction (Cox) technique will be used for 10 minutes. Developed in 1973, this chiropractic method uses a specialized table to decompress the spine, improve mobility, and reduce pain. Exercises include Pelvic Tilt, Hip Flexor Stretch, Hamstring Stretch, Cat-Camel, Bridge, and Straight Leg Raise, targeting flexibility, strength, and pain relief. Hot packs increase circulation and relax muscles. Both treatments are applied 3 times weekly for 4 weeks, ensuring consistent therapeutic benefits.
  Interventions: Other: mobilization

INTERVENTIONS:
Other: exercise — Ultrasound (4 minutes), TENS (100 Hz, 20 minutes), heat application (15 minutes), and home exercises will be applied. Treatment will be conducted three times a week for four weeks.
  Arms: Conventional Physical Therapy Group (CPTG)
Other: mobilization — In addition to heat application (15 minutes) and home exercises, the Cox technique will be used. The patient will be placed face down on a specialized table, and traction will be applied to the lumbar spine for 10 minutes.
  Arms: Flexion-Distraction Group (Cox Technique) (CTG):

SUMMARY:
The aim of this study is to compare the effects of conventional physical therapy and flexion-distraction (Cox technique) on pain, functional capacity, and quality of life in patients with lumbar disc herniation (LDH) receiving non-surgical treatment. The study will include two groups: one group will receive conventional physical therapy (ultrasound, transcutaneous electrical nerve stimulation (TENS), heat application, and home exercises), while the other group will receive heat application, the Cox technique, and home exercises. The effectiveness of these two methods will be compared to determine the most appropriate approach for LDH treatment.

The study will include individuals aged 30-60 diagnosed with L4-L5 disc herniation who apply to the Physical Medicine and Rehabilitation Department of Bursa VM Medical Park Hospital and Nilüfer Spine Health Center. Two groups of 34 participants each will be formed, and randomization will be based on the participants' preferred treatment center. The groups will be named the conventional physical therapy group (CPTG) and the Cox technique treatment group (CTTG).

Assessment parameters will include pain (visual analog scale (VAS) and algometry), range of motion (digital goniometer), functional capacity (Oswestry Disability Index - ODI), and quality of life (SF-36 Quality of Life Scale). Evaluations will be conducted by the same expert physiotherapist.

The treatment protocols are as follows:

Conventional Physical Therapy Group (CPTG): Ultrasound (4 minutes), TENS (100 Hz, 20 minutes), heat application (15 minutes), and home exercises will be applied. Treatment will be conducted three times a week for four weeks.

Flexion-Distraction Group (Cox Technique) (CTTG): In addition to heat application (15 minutes) and home exercises, the Cox technique will be used. The patient will be placed face down on a specialized table, and traction will be applied to the lumbar spine for 10 minutes.

Both groups will perform pelvic tilt, hip flexor stretching, hamstring stretching, cat-camel, bridge, and straight leg raise exercises, each repeated ten times.

The sample size was determined based on a study by Martinez et al., and a total of 68 participants will be included. Power analysis using the G*Power 3.1 program calculated the minimum sample size as 68.

Data will be analyzed using SPSS 25.0 software. Normal distribution will be evaluated using the Kolmogorov-Smirnov and Shapiro-Wilk tests. Parametric or non-parametric tests will be applied accordingly. Differences between groups will be analyzed using an independent samples t-test or the Mann-Whitney U test. Correlation analyses will be performed using Pearson or Spearman methods, and regression analyses will be applied to examine variable relationships.

The results of this study will contribute to determining the most effective conservative treatment approach for LDH patients by comparing the effectiveness of conventional physical therapy and the Cox technique.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of conventional physical therapy and flexion-distraction (Cox technique) on pain, functional capacity, and quality of life in patients with lumbar disc herniation (LDH) receiving non-surgical treatment. One group will receive conventional physical therapy (ultrasound, transcutaneous electrical nerve stimulation (TENS), heat application, and home exercises), while the other group will receive heat application, the Cox technique, and home exercises. The effectiveness of these two methods will be evaluated to determine the most appropriate approach for LDH treatment.

LDH is a condition in which damage to the disc structures compresses the nerve roots, causing pain, numbness, and movement limitations in the lower back and legs. Non-surgical methods are generally the first choice in treatment and have shown successful results. Conventional physical therapy methods are effective in pain management and functional improvement and are widely used to reduce muscle spasms and inflammation. Ultrasound provides thermal and mechanical effects on deep tissues, while TENS stimulates nerves to relieve pain. Heat application helps muscle relaxation and increases blood circulation.

Flexion-distraction (Cox technique) is a manual therapy method that aims to widen the spinal canal and reduce nerve compression. This technique increases the flexibility of spinal segments, alleviating pain and improving functional capacity. Randomized controlled studies have shown that this method is effective in LDH patients. However, studies directly comparing the Cox technique with conventional physical therapy are limited.

This study will include individuals aged 30-60 diagnosed with L4-L5 disc herniation who apply to the Physical Medicine and Rehabilitation Department of Bursa VM Medical Park Hospital and Nilüfer Spine Health Center. Two groups of 34 participants each will be included, and randomization will be based on the participants' preferred treatment center. The groups will be named the conventional physical therapy group (CTG) and the Cox technique treatment group (CTG).

Assessment parameters will include pain measurement using the visual analog scale (VAS) and algometry. Range of motion will be determined using a digital goniometer, functional capacity will be assessed with the Oswestry Disability Index (ODI), and quality of life will be measured with the SF-36 Quality of Life Scale. Evaluations will be conducted by the same expert physiotherapist.

The treatment protocols are as follows:

1. Conventional Physical Therapy Group (CTG): Ultrasound (4 minutes), TENS (100 Hz, 20 minutes), heat application (15 minutes), and home exercises will be applied. Treatment will be conducted three times a week for four weeks.
2. Flexion-Distraction Group (Cox Technique) (CTG): In addition to heat application (15 minutes) and home exercises, the Cox technique will be used. The patient will be placed face down on a specialized table, and traction will be applied to the lumbar spine for 10 minutes.

Both groups will perform pelvic tilt, hip flexor stretching, hamstring stretching, cat-camel, bridge, and straight leg raise exercises, each repeated ten times.

The sample size was determined based on a study by Martinez et al., and a total of 68 participants will be included. Power analysis using the G*Power 3.1 program calculated the minimum sample size as 68.

Data will be analyzed using SPSS 25.0 software. Normal distribution will be evaluated using the Kolmogorov-Smirnov and Shapiro-Wilk tests. Parametric tests will be used for normally distributed data, while non-parametric tests will be applied otherwise. Differences between groups will be analyzed using an independent samples t-test or the Mann-Whitney U test. Correlation analyses will be performed using Pearson or Spearman methods, and regression analyses will be applied to examine variable relationships.

The results of this study will contribute to determining the most effective conservative treatment approach for LDH patients by comparing the effectiveness of conventional physical therapy and the Cox technique.

ELIGIBILITY:
Inclusion Criteria:

* Being between 30-60 years of age
* Having a diagnosis of L4-L5 lumbar disc herniation
* Not having undergone surgical intervention
* Having no cognitive impairment or intellectual disability
* Providing voluntary participation and written consent

Exclusion Criteria:

* Having previously undergone surgical operation in the lumbar region
* Having an oncological diagnosis
* Pregnancy
* Presence of severe physical or psychological disorders that would prevent completion of the study
* Participation in another active physical therapy program

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-04-02 (Estimated); Primary Completion 2026-04-03 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
subjective pain | through study completion, an average of 6 months
  Measurements will be taken in two ways:
  Visual Analog Scale (VAS):
  The VAS scale will be used to assess low back pain in individuals with LDH. Participants will mark their pain level on a 10 cm line, where 0 represents "no pain" and 10 represents "very severe pain".
range of motion | through study completion, an average of 6 months
  Measurements will be taken using the Baseline goniometer, a digital goniometer. A digital goniometer is a tool used to precisely measure the range of motion of joints. It offers greater accuracy compared to traditional goniometers and displays measurements on a digital screen. Research shows that measurements taken with a digital goniometer provide more consistent results compared to traditional methods. The flexion, extension, lateral flexion, and rotation degrees of the lumbar region will be measured.
objective pain | through study completion, an average of 6 months
  Algometer:
  Measurements will be taken using the Baseline dolorimeter, a device that applies pressure to measure pain threshold. The algometer determines the pressure point at which the patient feels pain, assessing pain tolerance and threshold. Measurements will be taken from the right and left sides of the affected spinal segment

SECONDARY OUTCOMES:
Functional capacity | through study completion, an average of 6 months
  Functional capacity will be evaluated using the Oswestry Disability Index (ODI). The ODI is a questionnaire scale designed to assess the impact of low back pain on daily life. It consists of 10 items, each scored from 0 to 5. The total score reflects the patient's functional capacity. The ODI is a widely used and highly valid scale for evaluating the functional status of patients with low back pain
Daily living activities | through study completion, an average of 6 months
  Daily living activities will be evaluated using the SF-36 Quality of Life Scale. The SF-36 is a questionnaire designed to assess individuals' overall health status and quality of life, covering both physical and mental health dimensions. It consists of 36 questions, and separate scores are calculated for each dimension. The SF-36 is widely used for quality of life assessment in various populations, and its reliability and validity have been well-established.